CLINICAL TRIAL: NCT00003653
Title: A Phase III Randomized Trial Comparing Intermittent Versus Continuous Androgen Suppression for Patients With Prostate-Specific-Antigen Progression in the Clinical Absence of Distant Metastases Following Radiotherapy for Prostate Cancer
Brief Title: Hormone Therapy in Treating Patients With Rising PSA Levels Following Radiation Therapy for Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR7; CAN-NCIC-PR7 (Other: PDQ); SWOG-JPR7 (Other: SWOG); ICR-CTSU-JPR7 (Other: CTSU); CDR0000066745 (Other: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Buserelin; Cyproterone Acetate; Flutamide; Goserelin; Leuprolide; nilutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Androgen Suppression (Active Comparator)
  Interventions: Drug: bicalutamide; Drug: buserelin; Drug: cyproterone acetate; Drug: flutamide; Drug: goserelin; Drug: leuprolide acetate; Drug: nilutamide
- Continuous Androgen Suppression (Active Comparator)
  Interventions: Drug: bicalutamide; Drug: buserelin; Drug: cyproterone acetate; Drug: flutamide; Drug: goserelin; Drug: leuprolide acetate; Drug: nilutamide

INTERVENTIONS:
Drug: bicalutamide — Patients on the IAS arm should receive a minimum of 4 weeks of antiandrogen and a total of 8 months of LHRH analog during each on-treatment interval. The dose and frequency of LHRH treatment will be determined by the drug being administered (Appendix IX). Patients on the IAS arm should not be given an LHRH analog injection at the end of month 8 unless the patient is transferred to continuous treatment as per protocol upon completion of the 8 month intermittent treatment.
  Patients may be treated with any commercially available LHRH analog and antiandrogen during or after protocol treatment (Appendix IX). Patients may switch drugs at any time during or after protocol treatment. The dose and schedule of treatment will depend on the agent used. Patients should continue to receive hormone therapy without interruption until hormone resistance has been documented
Drug: buserelin — Patients on the IAS arm should receive a minimum of 4 weeks of antiandrogen and a total of 8 months of LHRH analog during each on-treatment interval. The dose and frequency of LHRH treatment will be determined by the drug being administered (Appendix IX). Patients on the IAS arm should not be given an LHRH analog injection at the end of month 8 unless the patient is transferred to continuous treatment as per protocol upon completion of the 8 month intermittent treatment.
  Patients may be treated with any commercially available LHRH analog and antiandrogen during or after protocol treatment (Appendix IX). Patients may switch drugs at any time during or after protocol treatment. The dose and schedule of treatment will depend on the agent used. Patients should continue to receive hormone therapy without interruption until hormone resistance has been documented
Drug: cyproterone acetate — Patients on the IAS arm should receive a minimum of 4 weeks of antiandrogen and a total of 8 months of LHRH analog during each on-treatment interval. The dose and frequency of LHRH treatment will be determined by the drug being administered (Appendix IX). Patients on the IAS arm should not be given an LHRH analog injection at the end of month 8 unless the patient is transferred to continuous treatment as per protocol upon completion of the 8 month intermittent treatment.
  Patients may be treated with any commercially available LHRH analog and antiandrogen during or after protocol treatment (Appendix IX). Patients may switch drugs at any time during or after protocol treatment. The dose and schedule of treatment will depend on the agent used. Patients should continue to receive hormone therapy without interruption until hormone resistance has been documented
Drug: flutamide — Patients on the IAS arm should receive a minimum of 4 weeks of antiandrogen and a total of 8 months of LHRH analog during each on-treatment interval. The dose and frequency of LHRH treatment will be determined by the drug being administered (Appendix IX). Patients on the IAS arm should not be given an LHRH analog injection at the end of month 8 unless the patient is transferred to continuous treatment as per protocol upon completion of the 8 month intermittent treatment.
  Patients may be treated with any commercially available LHRH analog and antiandrogen during or after protocol treatment (Appendix IX). Patients may switch drugs at any time during or after protocol treatment. The dose and schedule of treatment will depend on the agent used. Patients should continue to receive hormone therapy without interruption until hormone resistance has been documented
Drug: goserelin — Patients on the IAS arm should receive a minimum of 4 weeks of antiandrogen and a total of 8 months of LHRH analog during each on-treatment interval. The dose and frequency of LHRH treatment will be determined by the drug being administered (Appendix IX). Patients on the IAS arm should not be given an LHRH analog injection at the end of month 8 unless the patient is transferred to continuous treatment as per protocol upon completion of the 8 month intermittent treatment.
  Patients may be treated with any commercially available LHRH analog and antiandrogen during or after protocol treatment (Appendix IX). Patients may switch drugs at any time during or after protocol treatment. The dose and schedule of treatment will depend on the agent used. Patients should continue to receive hormone therapy without interruption until hormone resistance has been documented
Drug: leuprolide acetate — Patients on the IAS arm should receive a minimum of 4 weeks of antiandrogen and a total of 8 months of LHRH analog during each on-treatment interval. The dose and frequency of LHRH treatment will be determined by the drug being administered (Appendix IX). Patients on the IAS arm should not be given an LHRH analog injection at the end of month 8 unless the patient is transferred to continuous treatment as per protocol upon completion of the 8 month intermittent treatment.
  Patients may be treated with any commercially available LHRH analog and antiandrogen during or after protocol treatment (Appendix IX). Patients may switch drugs at any time during or after protocol treatment. The dose and schedule of treatment will depend on the agent used. Patients should continue to receive hormone therapy without interruption until hormone resistance has been documented
Drug: nilutamide — Patients on the IAS arm should receive a minimum of 4 weeks of antiandrogen and a total of 8 months of LHRH analog during each on-treatment interval. The dose and frequency of LHRH treatment will be determined by the drug being administered (Appendix IX). Patients on the IAS arm should not be given an LHRH analog injection at the end of month 8 unless the patient is transferred to continuous treatment as per protocol upon completion of the 8 month intermittent treatment.
  Patients may be treated with any commercially available LHRH analog and antiandrogen during or after protocol treatment (Appendix IX). Patients may switch drugs at any time during or after protocol treatment. The dose and schedule of treatment will depend on the agent used. Patients should continue to receive hormone therapy without interruption until hormone resistance has been documented

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Hormone therapy may fight prostate cancer by reducing the production of androgens. It is not yet known which androgen suppression regimen is more effective for prostate cancer.

PURPOSE: This randomized phase III trial is studying two hormone therapy regimens and comparing them to see how well they work in treating patients with rising PSA levels following radiation therapy for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of prostate cancer patients with prostate-specific antigen progression in the clinical absence of distant metastases after prior radical radiotherapy treated with intermittent androgen suppression (IAS) vs continuous androgen deprivation (CAD).
* Compare the time to the development of hormone resistance in patients treated with these regimens.
* Compare the quality of life of patients treated with these regimens.
* Compare the serum cholesterol and HDL/LDL levels at 3 years with those at baseline and compare them annually in patients treated with these regimens.
* Evaluate the duration of treatment and non-treatment intervals, time to testosterone recovery (return to pre-therapy levels), and time to recover potency in patients treated with IAS.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior radical prostatectomy (yes vs no), time since completion of prior radical radiotherapy (1 to 3 years vs 3 years or more), baseline prostate-specific antigen (PSA) value (3-15 ng/mL vs greater than 15 ng/mL), and prior hormonal therapy (neo-adjuvant, concurrent, or adjuvant cytoreduction in association with the radical radiotherapy treatment or prostatectomy for a maximum duration of 12 months and completed at least 12 months prior to randomization) (yes vs no). Patients are randomized to one of two treatment arms.

* Arm I: Patients undergo intermittent androgen suppression (IAS). Patients receive luteinizing hormone-releasing hormone (LHRH) analog (buserelin [BSRL], goserelin [ZDX], or leuprolide [LEUP]) and an antiandrogen (nilutamide [ANAN], flutamide [FLUT], bicalutamide [CDX], or cyproterone acetate [CPTR]) for 8 months. Patients receive LHRH analog by subcutaneous (SC) or intramuscular (IM) implant every 1-4 months beginning within 5 days of randomization and oral antiandrogen 1-3 times daily, depending on the actual LHRH analog and antiandrogen. PSA levels are monitored every 2 months. If PSA falls to normal during the 8-month treatment period, therapy stops until levels rise to 10 ng/mL, at which time IAS resumes for another 8-month period. IAS continues as long as PSA levels are controlled. At the time of disease progression, patients begin continuous hormonal treatment similar to arm II.
* Arm II: Patients undergo continuous androgen deprivation without scheduled interruptions. Patients receive LHRH analog (BSRL, ZDX, or LEUP) with an antiandrogen (ANAN, FLUT, CDX, or CPTR) OR undergo bilateral orchiectomy within 5 days of randomization and receive an antiandrogen. Patients receive LHRH analog by SC or IM implant every 1-4 months beginning within 5 days of randomization and oral antiandrogen 1-3 times daily, depending on the actual LHRH analog and antiandrogen. PSA levels are monitored every 2 months. Treatment continues until hormone resistance develops.

Patients receiving LHRH analog may begin antiandrogen therapy either prior to or simultaneously with LHRH analog and must continue antiandrogen therapy for at least 4 weeks to block tumor flare.

Quality of life is assessed at randomization, every 4 months for 2 years, every 8 months until development of hormone resistance, at the time of hormone resistance, and then annually thereafter.

Patients are followed annually for survival.

PROJECTED ACCRUAL: A total of 1,386 patients will be accrued for this study within 7 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven adenocarcinoma of the prostate prior to the initiation of radiotherapy
* Prior pelvic radiotherapy for prostate cancer, either post-radical prostatectomy or as primary management

  * More than 30 months since prior brachytherapy with curative intent
* Prostate-specific antigen must be rising and greater than 3 ng/mL and higher than the lowest level recorded previously since the end of radiotherapy (i.e., higher than the post-radiotherapy nadir)
* Total testosterone greater than 5 nmol/L
* No definite evidence of metastatic disease

  * Chest x-ray and bone scan negative for metastases
  * Radiological changes compatible with nonmalignant diseases allowed
* Clinical evidence of local disease allowed

PATIENT CHARACTERISTICS:

Age:

* 16 and over (18 and over for participating centers in the United Kingdom)

Performance status:

* ECOG 0-1

Life expectancy:

* More than 5 years

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 1.5 times ULN
* LDH no greater than 1.5 times ULN
* No chronic liver disease

Renal:

* Creatinine no greater than 1.5 times ULN

Other:

* Sufficiently fluent and willing to complete the quality of life questionnaire in either English or French
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except curatively treated basal or squamous cell skin cancer or superficial bladder cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior or concurrent biologic therapy

Chemotherapy:

* No prior or concurrent chemotherapy

Endocrine therapy:

* Prior hormonal therapy administered prior to, during, or immediately after radical radiotherapy or prostatectomy allowed provided duration was no longer than 12 months

  * At least 12 months since prior hormonal therapy

Radiotherapy:

* See Disease Characteristics
* At least 12 months since prior radiotherapy
* No concurrent palliative radiotherapy

Surgery:

* See Disease Characteristics
* See Endocrine therapy

Other:

* No concurrent bisphosphonates

Ages: 16 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1386 (Actual)
Dates: Start 1999-01-05 (Actual); Primary Completion 2010-10-04 (Actual); Study Completion 2013-01-10 (Actual)

PRIMARY OUTCOMES:
Overall survival | 2 years

SECONDARY OUTCOMES:
Time to hormone resistance | 2 years
Quality of life by European Organization for Research of the Treatment of Cancer Quality of Life Questionnaire-C30+ (EORTC QLQ-C30+) trial specific checklist | 2 years
Serum cholesterol, high-density lipoprotein, and low-density lipoprotein levels | 2 years
Duration of treatment and non-treatment interval during intermittent androgen suppression arm only | 2 years
Time to testosterone recovery during intermittent androgen suppression arm only | 2 years
Time to recovery of potency during intermittent androgen suppression arm only | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurence H. Klotz, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre; Celestia S. Higano, MD, Study Chair — University of Washington
Locations (29):
- Canada (29):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Fraser Valley Cancer Centre, Surrey, British Columbia
  - Clinical Research Unit at Vancouver Coastal, Vancouver, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - The Vitalite Health Network - Dr. Leon Richard, Moncton, New Brunswick
  - Atlantic Health Sciences Corporation, Saint John, New Brunswick
  - Dr. H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Center, Halifax, Nova Scotia
  - William Osler Health Centre, Brampton Memorial, Brampton, Ontario
  - Northeast Cancer Center Health Sciences, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Health Research Institute - General Division, Ottawa, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CHUM - Hopital Notre-Dame, Montreal, Quebec
  - McGill University - Dept. Oncology, Montreal, Quebec
  - CHUQ-Pavillon Hotel-Dieu de Quebec, Québec, Quebec
  - Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klotz L, Correia A, Zhang W. The relationship between the androgen receptor CAG repeat polymorphism length and the response to intermittent androgen suppression therapy for advanced prostate cancer. Prostate Cancer Prostatic Dis. 2005;8(2):179-83. doi: 10.1038/sj.pcan.4500792. PMID 15809670
- [Result] Crook JM, O'Callaghan CJ, Duncan G, Dearnaley DP, Higano CS, Horwitz EM, Frymire E, Malone S, Chin J, Nabid A, Warde P, Corbett T, Angyalfi S, Goldenberg SL, Gospodarowicz MK, Saad F, Logue JP, Hall E, Schellhammer PF, Ding K, Klotz L. Intermittent androgen suppression for rising PSA level after radiotherapy. N Engl J Med. 2012 Sep 6;367(10):895-903. doi: 10.1056/NEJMoa1201546. PMID 22931259
- [Derived] Hamilton RJ, Ding K, Crook JM, O'Callaghan CJ, Higano CS, Dearnaley DP, Horwitz EM, Goldenberg SL, Gospodarowicz MK, Klotz L. The Association Between Statin Use and Outcomes in Patients Initiating Androgen Deprivation Therapy. Eur Urol. 2021 Apr;79(4):446-452. doi: 10.1016/j.eururo.2020.12.031. Epub 2020 Dec 31. PMID 33390282
- [Derived] Klotz L, O'Callaghan C, Ding K, Toren P, Dearnaley D, Higano CS, Horwitz E, Malone S, Goldenberg L, Gospodarowicz M, Crook JM. Nadir testosterone within first year of androgen-deprivation therapy (ADT) predicts for time to castration-resistant progression: a secondary analysis of the PR-7 trial of intermittent versus continuous ADT. J Clin Oncol. 2015 Apr 1;33(10):1151-6. doi: 10.1200/JCO.2014.58.2973. Epub 2015 Mar 2. PMID 25732157